CLINICAL TRIAL: NCT02803281
Title: Assessment of Patient Frailty Prior to Thoracic Surgery: A Feasibility Study
Brief Title: Assessment of Patient Frailty Prior to Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 15-9170
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer; Esophageal Cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung Cancer - Frialty Assessment: Patients who will undergo surgery for lung cancer
  Interventions: Other: Frailty Assessment
- Esophageal Cancer - Frailty Assessment: Patients who will undergo esophagectomy for esophageal cancer
  Interventions: Other: Frailty Assessment

INTERVENTIONS:
Other: Frailty Assessment — Various physiologic and frailty assessment tests

SUMMARY:
Determine the feasibility of assessment of measures of frailty and determine if these measures provide a clinically important contribution of risk assessment in a population of patients undergoing major thoracic surgery for lung or esophageal cancer.

DETAILED DESCRIPTION:
Both gastro-esophageal and lung cancers are major causes of morbidity and mortality worldwide. In Canada the incidence for Esophageal Adenocarcinoma has doubled in the last two decades, while lung cancer is the leading cause of cancer death. Surgery is a treatment option for these patients; however, esophagectomy in particular, is associated with significant morbidity, mortality and adverse effect on quality of life. Despite satisfactory standard preoperative testing to evaluate risk for surgery, some patients experience morbidity and never recover fully from surgery. Frailty assessment may offer a more sensitive measure of a patient's physiologic reserve, which may allow identification of patients who are poor candidates for surgery. There is a lack of consensus of how best to assess frailty prior to surgery. This study aims to analyze frailty assessment as a tool for patient selection for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Esophageal or Lung Cancer who will undergo resectional surgery.

Exclusion Criteria:

* Patients undergoing diagnostic or staging procedures or pulmonary wedge excisions will be excluded.
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Patients - Lung or Esophageal
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Feasibility Assessment | 2 years
  Determine the feasibility of assessment of measures of frailty and determine if these measures provide a clinically important contribution of risk assessment in a population of patients undergoing major thoracic surgery for lung or esophageal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Gail E Darling, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - University Health Network (Toronto General Hospital), Toronto, Ontario
  - University Health Network: Toronto General Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Background] Hodari A, Hammoud ZT, Borgi JF, Tsiouris A, Rubinfeld IS. Assessment of morbidity and mortality after esophagectomy using a modified frailty index. Ann Thorac Surg. 2013 Oct;96(4):1240-1245. doi: 10.1016/j.athoracsur.2013.05.051. Epub 2013 Jul 31. PMID 23915593
- [Background] Talsma AK, Damhuis RA, Steyerberg EW, Rosman C, van Lanschot JJ, Wijnhoven BP. Determinants of improved survival after oesophagectomy for cancer. Br J Surg. 2015 May;102(6):668-75. doi: 10.1002/bjs.9792. Epub 2015 Mar 18. PMID 25787705
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Robinson TN, Eiseman B, Wallace JI, Church SD, McFann KK, Pfister SM, Sharp TJ, Moss M. Redefining geriatric preoperative assessment using frailty, disability and co-morbidity. Ann Surg. 2009 Sep;250(3):449-55. doi: 10.1097/SLA.0b013e3181b45598. PMID 19730176
- [Background] Chen CH, Ho-Chang, Huang YZ, Hung TT. Hand-grip strength is a simple and effective outcome predictor in esophageal cancer following esophagectomy with reconstruction: a prospective study. J Cardiothorac Surg. 2011 Aug 15;6:98. doi: 10.1186/1749-8090-6-98. PMID 21843340
- [Background] Yano Y, Inokuchi T, Kario K. Walking speed is a useful marker of frailty in older persons. JAMA Intern Med. 2013 Feb 25;173(4):325-6. doi: 10.1001/jamainternmed.2013.1629. No abstract available. PMID 23440240
- [Background] Fritz S, Lusardi M. White paper: "walking speed: the sixth vital sign". J Geriatr Phys Ther. 2009;32(2):46-9. No abstract available. PMID 20039582
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Sheetz KH, Zhao L, Holcombe SA, Wang SC, Reddy RM, Lin J, Orringer MB, Chang AC. Decreased core muscle size is associated with worse patient survival following esophagectomy for cancer. Dis Esophagus. 2013 Sep-Oct;26(7):716-22. doi: 10.1111/dote.12020. Epub 2013 Jan 25. PMID 23350746
- [Background] Rogalla P, Meiri N, Hoksch B, Boeing H, Hamm B. Low-dose spiral computed tomography for measuring abdominal fat volume and distribution in a clinical setting. Eur J Clin Nutr. 1998 Aug;52(8):597-602. doi: 10.1038/sj.ejcn.1600612. PMID 9725661
- See also: Canadian Cancer Statistics 2010 — http://www.cancer.ca